CLINICAL TRIAL: NCT05235815
Title: Ultrasound-Guided Retro Superior Costotransverse Ligament (SCTL) Compartment Block: Description of Sonoanatomy, Technique and Block Dynamics
Brief Title: Ultrasound- Guided Retro Superior Costotransverse Ligament (SCTL) Compartment Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Retro SCTL Block ver3
Record Dates: First submitted 2022-01-20; First posted 2022-02-11 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Thoracic Surgery, Video-Assisted
Keywords: Superior costotransverse ligament; Video assisted thoracoscopic surgery; Thoracic paravertebral block; Retro superior costotransverse ligament compartment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonoanatomy and retro SCTL compartment block (Experimental): During phase 1, ten healthy human volunteers will be involved. A bilateral ultrasound scan will be performed in the paravertebral region to describe the sonoanatomy of the retro SCTL compartment.
  During phase 2, participants who are scheduled for video-assisted thoracoscopic surgery (VATS) will receive an ultrasound-guided multi-level (T3-4, T5-6 and T7-8) retro SCTL compartment block.
  Interventions: Procedure: Retro SCTL compartment block

INTERVENTIONS:
Procedure: Retro SCTL compartment block — For phase 1, healthy human volunteers will be positioned in the lateral position with the side to be scanned in the non-dependent position. An ultrasound scan sequence to describe the retro SCTL space will be performed on both sides.
  During phase 2, participants who are scheduled for video-assisted thoracoscopic surgery (VATS) will receive an ultrasound-guided multi-level (T3-4, T5-6 and T7-8) retro SCTL compartment block. After positioning the participants, cleaning and draping the injection site, under sterile aseptic precautions and local anaesthetic infiltration, the block needle is inserted at the corresponding vertebral level (T7-T8) under ultrasound guidance in-plane to the ultrasound beam. Once the needle tip reaches the lateral aspect of the inferior articular process and behind the SCTL ligament, the desired volume (6ml/each level) of LA will be injected. This process will be continued at the remaining two vertebral levels (T5-T6 and T3-T4).

SUMMARY:
Thoracic paravertebral block (TPVB) is a regional anaesthetic technique that produces ipsilateral, segmental, somatic and sympathetic nerve blockade of multiple contiguous thoracic dermatomes. Although it is a safe technique, the needle tip comes close to the pleura during the injection, therefore, increasing the potential for pleural puncture and pneumothorax, especially when performed by inexperienced physicians. With the recently described retro superior costotransverse ligament (SCTL) compartment (using MRI) which has been shown to be in direct continuity with the intervertebral foramen, the investigators propose that the block needle need not pierce the SCTL and lie close to the pleura but can be positioned safely behind the ligament to deposit the local anaesthetic (LA). Therefore, this study aims to describe the sonoanatomy of the retro SCTL compartment and evaluate the block injection technique and sensory dynamics in patients scheduled for video-assisted thoracoscopic surgery (VATS).

DETAILED DESCRIPTION:
During a TPVB the LA is injected into the paravertebral space adjacent to the thoracic vertebra and close to the intervertebral foramen. Traditionally, either landmark or ultrasound-guided, TPVB is performed by depositing the LA anterior to the superior costotransverse ligament (SCTL), i.e. the block needle typically pierces the SCTL to reach the wedge-shaped TPVB space. Although it is a safe technique, the needle tip comes close to the pleura during the injection, therefore, increasing the potential for pleural puncture and pneumothorax, especially when performed by inexperienced physicians.

Recently, with the help of 3D micro computer tomography (CT), Cho T and colleagues have demonstrated in cadavers that the medial part of the SCTL does not end at the base of the transverse process but extends anteriorly to the vertebral body dividing the wedge-shaped paravertebral space into a retro SCTL compartment (posterior to SCTL) and a true paravertebral space (anterior to SCTL). Also, they demonstrated that the SCTL, as it extends to the vertebral body, forms a medial slit near the intervertebral foramen through which the ventral rami enters the true paravertebral space. Furthermore, they highlighted that the retro SCTL space or compartment is in direct communication with the intervertebral foramen and epidural space medially and to the true paravertebral space (through the medial and lateral slits). It is evident from their study that the retro SCTL compartment contains both the divisions of the spinal nerve, i.e., the ventral and dorsal rami, the latter exits the compartment to enter the erector spinae plane. Hence, with this new concept, it appears that the block needle tip needs not to pierce the SCTL as required in a conventional TPVB and LA deposited at the retro SCTL compartment, theoretically can spread to the paravertebral space, intervertebral foramen and the epidural space, to block the spinal nerves and its divisions, and the sympathetic trunks. The investigators believe that the LA injection in the retro SCTL compartment, owing to its close relationship with the intervertebral foramen, thoracic spinal nerve, and the sympathetic trunks, will also produce rapid onset of ipsilateral and or bilateral segmental somatic and sympathetic blockade of the thoracic dermatomes, akin to TPVB. In addition, as the needle tip lies farther away from the pleura (posterior to SCTL) the investigators believe that this technique may also be safer in terms of the potential risk of pleural puncture or pneumothorax than a conventional TPVB.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1: Healthy volunteers of age 18-60 years
* Phase 2: Patients age 18-80 years scheduled for video assisted thoracoscopic surgery (VATS)

Exclusion Criteria:

* Phase 2: 1. Patient refusal 2. Local skin site infection 3. Coagulopathy 4. History of allergy to local anesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Ultrasound visualization of the retro SCTL compartment in volunteers | Within 30 minutes after entering the procedure room
  The following structures will be assessed:
  1. The SCTL,
  2. The medial extension of SCTL in front of the intervertebral foramen,
  3. The retro SCTL compartment behind the medial extension of the SCTL, and
  4. The true paravertebral space.
  The quality of ultrasound visibility (ultrasound visibility score, UVS) of each structure will be assessed using a 4-point Likert scale (0= not visible, 1= hardly visible, 2= well visible, 3= very well visible).
Readiness for surgery | Within 30 minutes after the block at 5 minutes interval
  An overall sensory score of =<30 on the ipsilateral hemithorax (loss of sensation to cold stimulus (ice cube), NRS: 0-100, 0= no sensation, 100= normal sensation)
  Sensation block assessment: T2-L5 spinal nerves

SECONDARY OUTCOMES:
Complete sensory block | Within 30 minutes after the block at 5 minutes interval
  An overall sensory score 0 on the ipsilateral hemithorax (loss of sensation to cold stimulus (ice cube), NRS: 0-100, 0= no sensation, 100= normal sensation)
  Sensation block assessment: T2-L5 spinal nerves
Block performance time | Within 30 minutes after entering the procedure room
  The time taken from the start of the local anaesthetic (LA) skin infiltration to the end of the LA injection for the block.
Total amount of vasopressor used | After completion of the block and through the surgical period, an average of 6 hours
  The total amount of vasopressor requirements after the completion of the block and through the surgical period will be recorded.
Total amount of morphine used | During surgical period and postanesthesia care unit (PACU) period, an average of 6 hours
  The total amount of morphine requirements through the surgical period and post anaesthesia care unit (PACU) period, until the discharge of participants from the PACU, will be recorded.
Postoperative pain score | At arrival and discharge from postanesthesia care unit (PACU)
  Postoperative pain score in the form of a numerical rating scale (NRS) will be recorded in the post anaesthesia care unit (PACU) at rest and movement (cough), at arrival and discharge from PACU.
  (NRS: 0-100, 0= no pain, 100= worst imaginable pain)
Postoperative sensory score before discharge | At discharge from postanesthesia care unit (PACU)
  Sensory score on bilateral hemithorax (loss of sensation to a cold stimulus (ice cube), NRS: 0-100, 0= no sensation, 100= normal sensation), when discharge from postanesthesia care unit (PACU).
  Sensation block assessment: T2-L5 spinal nerves
Complications | Within 45 minutes after the block, within 24 hours post surgery and at 1 week after the surgery
  Any complication directly related to the retro SCTL compartment block (vascular puncture, pleural puncture, or local anaesthetic toxicity) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong